CLINICAL TRIAL: NCT01750099
Title: A Randomized Single-blinded Trial of Combined Spinal-Epidural Versus Continuous Epidural Analgesia
Brief Title: Pain Relief Effects on Length of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Erica Grant, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 042012-035
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Labor Pain
Keywords: Labor; analgesia; epidural; spinal
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Fentanyl; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined spinal-epidural (Experimental): After verification of being in the intrathecal space with free-flow of cerebral spinal fluid, 1 mL of 0.25% bupivicaine along with 20 mcg of fentanyl will be injected into the intrathecal space. Subsequently, a B/Braun Perifix FX closed tip multiorifice flexible epidural catheter will be threaded 4 cm into the epidural space. After obtaining a T6 dermatomal level of sensory blockade, a standard solution consisting of 0.125% bupivicaine with 2 mcg of fentanyl/mL of solution will be started at 10 mL/hour with a patient controlled epidural analgesia (PCEA) option of 8 mL every 45 minutes. If a patient requires redosing, 5-10 mL of 0.25% bupivicaine will be injected slowly through epidural catheter with a goal dermatome level of T6. No systemic opioids will be given.
  Interventions: Procedure: Combined Spinal-epidural
- Continuous lumbar epidural (Placebo Comparator): After identifying the epidural space with the loss of resistance technique, a standard flexible epidural catheter will be threaded 4 cm into the epidural space. A standard test dose of 3 mL of 1.5% lidocaine with epinephrine 1:200,000 will be given through the catheter. If positive for vascular or intrathecal placement, procedure to be repeated at different interspace. If negative, catheter will be secured and slowly dosed with 5-10 mL of 0.25% bupivicaine through epidural catheter with a goal dermatome level of T6. After obtaining the dermatome level of sensory blockade, a standard solution consisting of 0.125% bupivicaine with 2 mcg of fentanyl/mL of solution will be started at 10 mL/hour with a PCEA option of 8 mL every 45 minutes. If a patient requires redosing, 5-10 mL of 0.25% bupivicaine will be injected slowly through epidural catheter with a goal dermatome level of T6. No systemic opioids will be given.
  Interventions: Procedure: Continuous Lumbar epidural

INTERVENTIONS:
Procedure: Combined Spinal-epidural — See arm description
  Other Names: Spinal dose: 1 ml of 0.25 % bupivicaine; 20 mcg of fentanyl; Epidural dose: 0.25 % bupivicaine (various amounts according to protocol); fentanyl
  Arms: Combined spinal-epidural
Procedure: Continuous Lumbar epidural — See arm description
  Other Names: 3 ml of 1.5% lidocaine with epinephrine 1:200000; 0.25 % bupivicaine; fentanyl
  Arms: Continuous lumbar epidural

SUMMARY:
This study divides patients into two groups when they ask for medicine to help relieve the pain of contractions. One group will be selected to receive an epidural and another group will be selected to receive both a spinal dose and an epidural. The investigators will then measure how long it takes to deliver the baby. The investigators think that the group that has the combination spinal and epidural will have a faster labor.

DETAILED DESCRIPTION:
In this randomized controlled trial, the investigators will evaluate conventional continuous lumbar epidural analgesia compared to the combined spinal-epidural analgesia. The primary outcome of interest will be duration of the active phase of the first stage of labor. Secondary outcomes include the cesarean delivery rate, operative vaginal delivery rate, analgesia requirements, maternal and neonatal safety profiles (incidence of maternal hypotension, post puncture dural headache, fetal acidemia and NICU admissions, respectively), Adequacy of maternal pain relief will also be measured using visual analog scores (VAS). The investigators hypothesize that the instantaneous pain relief that is achieved with combined spinal-epidural analgesia reduces catecholamines quickly and to a greater degree than the conventional epidural, leading to a more effective uterine contraction pattern thus decreasing the duration of the active phase of the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Term gestation, defined as equal to or greater than 37 weeks
* Ages 16-44 years
* Singleton gestation
* Cephalic presentation
* Induction of labor on Monday 0700 through Friday 0700 at Parkland Hospital
* Intact membranes on admission

Exclusion Criteria:

* Chorioamnionitis at randomization
* Intrauterine fetal death
* Coagulopathy
* Allergies to amide local anesthetics
* Localized back infection

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 202 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Duration of stage I labor | 1.5 years

SECONDARY OUTCOMES:
Incidence of operative vaginal delivery | 1.5 years

OTHER OUTCOMES:
Incidence of cesarean delivery rate | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Erica N Grant, MD, Principal Investigator — UTSW; Kenneth Leveno, MD, Study Director — UTSW
Locations (1):
- Parkland Hospital, Dallas, Texas, United States